CLINICAL TRIAL: NCT05649033
Title: Work-related Stress Among Recently Graduated Midwives Practicing in the Delivery Room
Acronym: Stress-SF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_009_Stress-SF
Record Dates: First submitted 2022-12-02; First posted 2022-12-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Recently Graduated Midwives Practicing in the Delivery Room
Keywords: midwives; Work-related stress; delivery room
MeSH Terms: conditions — Occupational Stress | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group "recently graduated midwives practicing in the delivery room": Midwives graduated for less than three years and practicing in the delivery room
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Work-related stress evaluation

SUMMARY:
Work stress results from an imbalance between the worker's hopes and work's conditions.

Midwifes are exposed to emergency situations (newborn distress, neonatal resuscitation, foetal abnormal heart rythm, delivery hemorrhage, …), which can cause stress and sometimes lead to burnout.

DETAILED DESCRIPTION:
the aim of the study is to describe Work-related stress among recently graduated midwives practicing in the delivery room

ELIGIBILITY:
Inclusion Criteria:

* Midwives graduated for less than three years in France
* Practicing in the delivery room
* Whatever the duration of exercise in the delivery room
* Agreeing to participate in the study

Exclusion Criteria:

* No Agreeing to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Midwives graduated for less than three years practicing in the delivery room
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Work-related stress | Day 0
  Work-related stress evaluated using Perceived Stress Scale (PPS10). PPS10 includes 10 items evaluating the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month. Each item is coded from 1 to 4 points: never, almost never, sometimes, fairly often and very often. The overall score ranges from 0 to 40 points.

CONTACTS AND LOCATIONS:
Overall Officials: Le Tarnec Louise Anne, Dr, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (1):
- Université de Reims Champagne Ardenne, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided